CLINICAL TRIAL: NCT06008457
Title: Prospective Clinical Evaluation of the Labcorp COVID-19+Flu+RSV Test Home Collection Kit as Offered Commercially by Labcorp - A Registry Study
Brief Title: Evaluation of the Labcorp COVID-19+Flu+RSV Test Home Collection Kit
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-VIR-403
Record Dates: First submitted 2023-08-21; First posted 2023-08-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COVID-19 Respiratory Infection; Influenza A; Influenza Type B; RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Remnant swab samples from all subjects (positive and negative) and isolated viral DNA will be maintained for future related research. No human DNA will be maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Self-collection first: Subjects will self-collect an anterior nasal swab first
  Interventions: Device: Labcorp COVID-19+Flu+RSV Test Home Collection Kit
- HCP-collection first: Subjects will have their healthcare provider collect an anterior nasal swab first
  Interventions: Device: Labcorp COVID-19+Flu+RSV Test Home Collection Kit

INTERVENTIONS:
Device: Labcorp COVID-19+Flu+RSV Test Home Collection Kit — The self-collected Labcorp COVID-19+Flu+RSV Test Home Collection Kit results as generated by the commercially available Labcorp Seasonal Respiratory Virus RT-PCR Test will be compared to the HCP-collected results as generated by Labcorp R&D using the comparator assays.

SUMMARY:
To compare the results obtained by analysis of a self-collected anterior nasal (AN) swab as part of the Labcorp COVID-19+Flu+RSV Test Home Collection Kit to a healthcare provider (HCP)-collected AN swab in patients with symptoms of viral respiratory infection consistent with influenza A (Flu A), influenza B (Flu B), respiratory syncytial virus (RSV) and/or SARS-CoV-2 (C-19).

ELIGIBILITY:
Inclusion Criteria:

* presents with symptoms of viral respiratory infection consistent with Flu A, Flu B, RSV and/or C-19;
* Subject can read and understand written instructions in English; and
* Subject is able, in the professional opinion of the investigator, to provide up to 18.5mL of whole blood at the clinic visit. NOTE - the blood draw will be optional for subjects <12 years of age.

Exclusion Criteria:

* Subject is 14-17 years of age and their parent or legal guardian is unable to supervise the collection of the AN swab sample from the subject;
* Subject is <14 years of age and their parent or legal guardian refuses to collect the AN swab sample from the subject; or
* Previous participation in this protocol.

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients ≥2 years of age who present to the participating study clinics with symptoms of viral respiratory infection consistent with Flu A, Flu B, RSV and/or C-19 and who meet all study inclusion criteria and no exclusion criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Collection method comparison | 1 day
  To evaluate the concordance between the results of a self-collected AN swab specimen using the Labcorp COVID-19+Flu+RSV Test Home Collection Kit as analyzed by the Labcorp Seasonal Respiratory Virus RT-PCR Test and an HCP-collected AN swab as analyzed by the comparator assays in subjects presenting with symptoms of viral respiratory infection consistent with Flu A, Flu B, RSV and/or C-19.

SECONDARY OUTCOMES:
Whole blood specimen collection | 1 day
  The whole blood specimen collection is designed to support assay research and/or development and validation of blood-based virology assays.

CONTACTS AND LOCATIONS:
Overall Officials: Graham McLennan, MS, Study Director — Laboratory Corporation of America
Locations (1):
- Exer Urgent Care, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share data